CLINICAL TRIAL: NCT00676702
Title: A Single-Dose, Open-Label, Randomized, Crossover Study to Evaluate Intraduodenal Enzyme Delivery of PANCREASE MT in Subjects With Severe Exocrine Pancreatic Insufficiency
Brief Title: A Study of the Enzyme Activity and Safety of Pancrelipase in Patients With Severe Exocrine Pancreatic Insufficiency (EPI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Senior Director Clinical Research and Development, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Model: Crossover
Other Study IDs: CR014716; PNCRLPCYS1001
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-02

CONDITIONS: Exocrine Pancreatic Insufficiency; Pancreatitis, Chronic; Steatorrhea; Pancreatitis
Keywords: Pancrelipase; PANCREASE MT; Cross-Over Studies; Duodenum; Intestine, Small; Lipase; Amylases; Peptide Hydrolases; Intubation; Safety; Capsules
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Pancreatitis, Chronic; Steatorrhea; Pancreatitis; Cerebral Palsy | interventions — Ensure Plus; Pancrelipase

ARMS (2):
- 001 (Experimental): Pancrelipase in combination with Ensure Plus 3 pancrelipase MT 21 capsules containing a total of 63 000 USP units of lipase with a high-fat liquid meal of 500 ml of Ensure Plus.
  Interventions: Drug: Pancrelipase in combination with Ensure Plus
- 002 (Active Comparator): Ensure Plus A high-fat liquid meal of 500 ml of Ensure Plus
  Interventions: Dietary Supplement: Ensure Plus

INTERVENTIONS:
Dietary Supplement: Ensure Plus — A high-fat liquid meal of 500 ml of Ensure Plus
  Arms: 002
Drug: Pancrelipase in combination with Ensure Plus — 3 pancrelipase MT 21 capsules containing a total of 63,000 USP units of lipase with a high-fat liquid meal of 500 ml of Ensure Plus.
  Arms: 001

SUMMARY:
The purpose of the study is to evaluate the enzyme activity and safety of pancrelipase in patients with severe Exocrine Pancreatic Insufficiency (EPI)

DETAILED DESCRIPTION:
Pancrelipase, the active ingredient in pancrelipase microtablet (MT) 21 capsules, is a pancreatic enzyme preparation (PEP) for oral administration that aids in the digestion of fats, sugars and proteins. Approximately 20 men and women from 18 to 85 years of age will be enrolled in the study. Patients enrolled must have severe pancreatic insufficiency with steatorrhea (presence of fat in the stool as a result of insufficient fat absorption in the digestive track) due to severe exocrine pancreatic insufficiency (EPI), a condition when the body is unable to digest food because the body does not have digestive enzymes made by the pancreas to digest fats, sugars and proteins properly for normal nutritional needs. The study will last approximately 25 days and will consist of a screening phase that will take place within 21 days before an open-label (patient knows the identity of the treatment they are receiving) treatment phase that will consist of 2 treatment periods (each treatment period will be approximately 4 hours long), a 2-day washout period between treatment periods, and an end-of-study evaluation upon successful completion of the sample collection in treatment period 2. Study participants will arrive at the study center no later than 6 p.m. on the day before treatment period 1 and stay overnight at the study center until the end-of-study evaluation in treatment period 2 (approximately 5 days). During the study, patients may not consume food or beverages containing alcohol, must refrain from the use of any methylxanthine-containing products, (eg, chocolate bars or beverages, coffee, teas, or colas), must eat only the meals provided during the study while residing at the study center, and must refrain from jogging, strenuous exercise of all types, and sunbathing. At the screening visit, patients will be asked to sign an informed consent form indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study. Patients will then be asked to provide information regarding their medical history and will have a complete physical examination (including heart and respiration rate, blood pressure, temperature, height, and weight) performed. In addition, a blood sample (10 mL or approximately 2 teaspoons of blood) and a urine sample will be collected to assess the patient's general health. A urine pregnancy test will also be performed on women of childbearing age. If the patient is eligible to participate in the study, he/she will be asked to stop taking any existing pancreatic enzymes, prescription and nonprescription medications (including vitamins and herbal supplements) that could affect the stomach or intestines for 3 to 7 days before returning to the study center for treatment periods 1 and 2. During the study, patients will receive either Treatment A in Period 1 and Treatment B in Period 2; or Treatment B in Period 1 and Treatment A in Period 2. The day before (Day -1) of treatment period 1, patients will be randomly (by chance) assigned to 1 of 2 treatment sequences (Treatment A or Treatment B). Treatment A will consist only of a high-fat liquid meal (500 mL of Ensure Plus containing 22.9 g of fat). Treatment B will consist of 3 PANCREASE MT 21 capsules taken orally (by mouth) along with a high-fat liquid meal (500 mL of Ensure Plus containing 22.9 g of fat). Following an overnight fast (without eating) of at least 10 hours, patients will be intubated (ie, have a tube inserted through their nose into the small intestine [duodenum]) in order to collect samples of fluid from their stomach and intestine before and after treatment in treatment periods 1 and 2. In treatment period 1, patients will be given the study treatment (Treatment A or Treatment B) orally (by mouth) over a 20-25 minute period, followed by a 2-hour sample collection period. After the sample completion period, the intubation tube will be removed and patients will have a washout period of at least 48 hours where they will rest and not receive treatment. At the end of the washout period, patients will enter treatment period 2 and receive the second study treatment. Patient's may be required to stay overnight for observation after the completion of the sample collection in Period 2, otherwise, patients will be permitted to leave the study center on Day 1 of treatment period 2 following a physical examination and collection of blood and urine samples for safety assessments. The primary outcome in the study is to evaluate the pharmacokinetics (enzyme activity) of intraduodenal enzyme (lipase, amylase, and protease) delivery of a single dose of 3 pancrelipase MT 21 capsules in gastric and duodenal fluid samples collected from patients before treatment and at 15 minute intervals up to 2 hours after treatment on Day 1 during each treatment period. During the study, the safety and tolerability of study drug will be monitored from the time of screening (Day -21) through to the end of the study procedures performed on Day 1 of treatment period 2 by evaluating adverse events (side effects), results from clinical laboratory tests (serum chemistry, hematology, and urinalysis), vital signs (blood pressure, pulse, respiratory rate, and body temperature) measurements, and findings from physical examinations reported. Adverse events reported by patients were also monitored for up to 30 days following discharge from the study center. On Day 1 of the first treatment period, patients will receive Treatment A (a high-fat liquid meal of 500 ml of Ensure Plus) OR Treatment B (3 pancrelipase microtablet (MT) 21 capsules taken orally by mouth in addition to a high-fat liquid meal of 500 ml of Ensure Plus) ingested within 20-25 minutes. After a 2-day washout period, in the second treatment period, patients who received Treatment A in period 1 will receive Treatment B and patients who received Treatment B will receive Treatment A.

ELIGIBILITY:
Inclusion Criteria:

* Must have evidence of chronic pancreatitis or pancreatic insufficiency (steatorrhea) confirmed prior to screening
* Must be able to discontinue treatment with any pancreatic enzyme preparations (PEPs) within 72 hours before admission to the study center for the open-label phase to the end-of-study evaluations (a total of approximately 7 days)
* If a woman, must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control (eg, prescription oral contraceptives, contraceptive injections, intrauterine device, double barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study and have a negative urine pregnancy test at screening
* Must have signed an informed consent document indicating an understanding of the purpose and procedures required for the study and willingness to participate in the study

Exclusion Criteria:

* Current significant medical and/or mental disease including solid organ transplant, massive small bowel resection, or major gastrointestinal or pancreatic surgery that potentially affect the intestinal absorption and metabolism of fat (excluding severe pancreatic insufficiency with steatorrhea due to chronic pancreatitis or exocrine pancreatic insufficiency)
* History of or current acute pancreatitis or acute exacerbations of chronic pancreatic disease, or coagulopathy
* Use of any prescription that can influence gastrointestinal physiology or any nonprescription medication (including vitamins and herbal supplements) except for acetaminophen, oral contraceptives, and hormonal replacement therapy, and local numbing agents, short-acting benzodiazepines, metoclopramide used during the placement of the intubation tube for up to 3 to 7 days before admission to the study center
* Known allergy to the study drug, pork protein, or any of the excipients of the pancreatic enzyme formulation or to medications used during the placement of the intubation tube (ie, local numbing agents, short-acting benzodiazepines, metoclopramide)
* Unable to swallow solid, oral dosage forms whole with the aid of a liquid meal (participants may not chew, divide, dissolve, or crush the study drug) and/or tolerate gastroduodenal intubation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics (enzyme activity) of intraduodenal enzyme (lipase, amylase, and protease) delivery of a single dose of 3 pancrelipase MT 21 capsules in gastric and duodenal fluid samples collected from patients | Pretreatment and at 15 minute intervals up to 2 hours posttreatment on Day 1 during each treatment period.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of 3 pancrelipase MT 21 capsules containing a total of 63,000 USP units of lipase. | Time of screening (Day -21) through to the end of the study procedures performed on Day 1 of treatment period 2.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the enzyme activity and safety of pancrelipase in patients with severe Exocrine Pancreatic Insufficiency (EPI) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=777&filename=CR014716_CSR.pdf